CLINICAL TRIAL: NCT06220591
Title: Ultrasound-guided Selective Supraclavicular Nerve Block with Either Superior Trunk or Clavipectoral Fascial Plane Block for Clavicular Surgery
Brief Title: Comparing Local Anesthetic Techniques for Clavicular Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Clavicular anesthesia
Record Dates: First submitted 2023-12-27; First posted 2024-01-24 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Superior trunk group (Active Comparator): The patient will undergo selective supraclavicular nerve block, then will undergo block of superior trunk "The fifth & sixth cervical nerve roots" of the brachial plexus on the side of the affected clavicle.
  Interventions: Procedure: Superior trunk block
- Clavipectoral fascial plane group (Active Comparator): The patient will undergo selective supraclavicular nerve block, then will undergo clavipectoral fascial plane block on the lateral and medial ends of the affected clavicle.
  Interventions: Procedure: Clavipectoral fascial plane block

INTERVENTIONS:
Procedure: Superior trunk block — The patient will receive selective supraclavicular nerve block, then will undergo blockage of superior trunk "the fifth and sixth cervical nerves" of the brachial plexus. The operator will scan the supraclavicular nerve on the lateral border of the sternomastoid muscle. Local anesthetics mixture"3 cc" will be injected in 0.5 cc aliquots after negative aspiration to encircle the supraclavicular nerve. Then ultrasound probe will be moved to scan the superior trunk "the fifth and sixth cervical nerves" in the scalene groove.15 cc of local anesthetics mixture will be injected in 0.5 cc aliquots to encircle the fifth & sixth cervical nerve roots.
  Arms: Superior trunk group
Procedure: Clavipectoral fascial plane block — The patient will receive selective supraclavicular nerve block, then will undergo clavipectoral fascial plane block. The operator will scan the supraclavicular nerve on the lateral border of the sternomastoid muscle. Local anesthetics mixture"3 cc" will be injected in 0.5 cc aliquots after negative aspiration to encircle the supraclavicular nerve. The ultrasound probe will scan both the medial & lateral ends of the clavicle. Then Local anesthetics mixture"15 cc" will be injected in 0.5 cc aliquots after negative aspiration between the periosteum of the clavicle and the clavipectoral fascia. The same technique will be conducted on both the lateral and medial ends of the affected clavicle.
  Arms: Clavipectoral fascial plane group

SUMMARY:
Surgical fixation for acute clavicular fractures is increasingly preferred among orthopedic surgeons to improve healing and decrease the risk of malunion. Regional anesthesia for clavicular fractures allows rapid recovery, prolonged postoperative analgesia, and less opioid consumption, and so decreases the hospital stay. There is no consensus regarding the best regional anesthetic technique for surgical fixation for acute clavicular fractures. Selective supraclavicular nerve block combined with either superior trunk or clavipectoral fascial plane block is a promising regional anesthetic technique for midshaft clavicular surgeries.

DETAILED DESCRIPTION:
This study will assess if there is a difference in the quality of surgical anesthesia between selective supraclavicular nerve block combined with either superior trunk or clavipectoral fascial plane block for clavicular fractures. Aiming to achieve high-quality surgical anesthesia and postoperative analgesia for middle clavicular fracture surgeries with optimum hemodynamic stability and high patient and surgeon satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years old.
* Sex: both sexes.
* The American Society of Anesthesiologists (ASA) Physical status: ASA I & II.
* Body mass index (BMI): 18.5 - 24.9 kg/m2.
* Type of operations: surgical repair of the midshaft clavicular injuries.

Exclusion Criteria:

* Patient refusal.
* Known hypersensitivity to lidocaine or bupivacaine.
* Patients with respiratory insufficiency.
* Coagulation disorders or taking drugs affect surgical hemostasis.
* Patients with pre-existing neurological deficits
* Uncooperative patient or with altered mental status.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-01-27 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Time of the first rescue analgesic request by the patient postoperative. | 24 hours
  The patient will be asked to quantify postoperative pain using the visual analogue pain score as the following 0: no pain, and 10: maximum imaginable pain. Nalbuphine 4 mg will be administered intravenous as rescue analgesia if the visual analogue pain score ≥4. The time of the first rescue analgesic request will be recorded.

SECONDARY OUTCOMES:
Onset of sensory block. | 20 minutes
  From the end of block procedure to the of loss of pin prick sensation will be tested over the affected clavicle.
Ipsilateral diaphragmatic excursion affection. | 1 hour
  Ipsilateral diaphragmatic excursion will be assessed by M-mode ultrasound.
The Numerical Pain Rating Scale in the first 24 hours | 24 hours.
  On a scale of 0-10, the patient will be asked to quantify postoperative pain as the following 0: no pain, and 10: maximum imaginable pain.
The total opioid consumption in the first 24 hours | 24 hours.
  The total dose of intravenous nalbuphine in the first 24 hours postoperatively
Patient and surgeon satisfaction. | 24 hours
  Patient and surgeon satisfaction will be assessed using 7- point Likert-like verbal rating scale.
Any reported complications. | 24 hours.
  The possible side effects will be followed in the first 24 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Fahmy, MD, Principal Investigator — Lecturer of Anesthesia, Intensive Care & Pain management, Faculty of Medicine, Zagazig University
Locations (1):
- Zagazig university hospital, Zagazig, Al-Sharkia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Postacchini F, Gumina S, De Santis P, Albo F. Epidemiology of clavicle fractures. J Shoulder Elbow Surg. 2002 Sep-Oct;11(5):452-6. doi: 10.1067/mse.2002.126613. PMID 12378163
- [Background] Virtanen KJ, Malmivaara AO, Remes VM, Paavola MP. Operative and nonoperative treatment of clavicle fractures in adults. Acta Orthop. 2012 Feb;83(1):65-73. doi: 10.3109/17453674.2011.652884. Epub 2012 Jan 17. PMID 22248169
- [Background] Banerjee S, Acharya R, Sriramka B. Ultrasound-Guided Inter-scalene Brachial Plexus Block with Superficial Cervical Plexus Block Compared with General Anesthesia in Patients Undergoing Clavicular Surgery: A Comparative Analysis. Anesth Essays Res. 2019 Jan-Mar;13(1):149-154. doi: 10.4103/aer.AER_185_18. PMID 31031496
- [Background] Valdes-Vilches LF, Sanchez-del Aguila MJ. Anesthesia for clavicular fracture: selective supraclavicular nerve block is the key. Reg Anesth Pain Med. 2014 May-Jun;39(3):258-9. doi: 10.1097/AAP.0000000000000057. No abstract available. PMID 24747317
- [Background] Kang R, Jeong JS, Chin KJ, Yoo JC, Lee JH, Choi SJ, Gwak MS, Hahm TS, Ko JS. Superior Trunk Block Provides Noninferior Analgesia Compared with Interscalene Brachial Plexus Block in Arthroscopic Shoulder Surgery. Anesthesiology. 2019 Dec;131(6):1316-1326. doi: 10.1097/ALN.0000000000002919. PMID 31490292
- [Background] Goncalves D, Sousa CP, Graca R, Miguelez MP, Sampaio C. Clavipectoral Fascia Plane Block Combined With Superficial Cervical Plexus Block for the Removal of Osteosynthesis Material From Clavicle Fracture. Cureus. 2023 Aug 8;15(8):e43146. doi: 10.7759/cureus.43146. eCollection 2023 Aug. PMID 37692707